CLINICAL TRIAL: NCT02097303
Title: Open Label Phase Two Trial of Radium Ra 223 Dichloride With Concurrent Administration of Abiraterone Acetate Plus Prednisone in Symptomatic Castration-Resistant (Hormone-Refractory) Prostate Cancer Subjects With Bone Metastasis
Acronym: eRADicAte
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carolina Research Professionals, LLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRP-PCA-01 eRADicAte
Record Dates: First submitted 2014-03-21; First posted 2014-03-27 (Estimated); Results first posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Bone Metastasis; Symptomatic; Androgen Independent; Hormone Refractory; Castrate Resistant; AIPC; pre-chemotherapy; Post-chemotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Other): All subjects receive concurrent administration of Radium Ra223 Dichloride and Abiraterone Acetate plus Prednisone
  Interventions: Drug: Concurrent use of Radium Ra 223 dichloride and Abiraterone Acetate plus Prednisone

INTERVENTIONS:
Drug: Concurrent use of Radium Ra 223 dichloride and Abiraterone Acetate plus Prednisone — Radium Ra 223 dichloride - A targeted alpha particle-emitting pharmaceutical (a radiopharmaceutical drug) is a ready-to-use solution for intravenous injection containing the drug substance radium dichloride. The active moiety is the alpha particle emitting nuclide Ra-223, present as a divalent cation (223Ra2+) and Abiraterone Acetate - A CYP17 inhibitor, indicated in combination with prednisone for the treatment of subjects with metastatic castration-resistant prostate cancer. Administration of Abiraterone Acetate may result in mineralocorticoid-related adverse events (AEs), due to CYP17 inhibition. Therefore, Abiraterone Acetate is administered in combination with Prednisone to reduce the frequency of these AEs.
  Other Names: Xofigo; Zytiga

SUMMARY:
This is an open label study designed to examine the effects on concurrent administration of Radium Ra 223 dichloride and Abiraterone Acetate plus Prednisone in subjects with symptomatic castrate resistant prostate cancer and with bone metastases, in both the pre- and post- chemotherapy setting. Both medications are approved by the US Food and Drug Administration for this indication.

DETAILED DESCRIPTION:
Approximately 40 subjects will be enrolled to obtain 30 evaluable subjects. All subjects will receive Radium Ra 223 dichloride every 4 weeks for a total of 6 doses over 24 weeks and concurrent Abiraterone Acetate plus Prednisone for a minimum duration of 26 weeks.

Subjects will be evaluated 30 days after the last dose of Radium Ra 223 dichloride. All adverse events deemed to be study related will be followed until resolution. Including screening, the total duration of the study is 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects will conform to all of the inclusion criteria listed below:

1. Subject must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
2. Subject is willing and able to comply with the protocol, including all study visits and procedures.
3. Subject is a male, greater than 18 years at time of enrollment.
4. Life expectancy of at least 9 months.
5. Subject has histologically documented prostate cancer confirmed by a pathology report from a prostate biopsy or radical prostatectomy specimen.
6. Subject must:

   • have initiated a stable dose of daily Abiraterone Acetate plus Prednisone within 90 days of enrollment, or

   • plans to initiate a stable daily dose of Abiraterone plus Prednisone within 30 days of the first Radium Ra 223 dichloride treatment.
7. Subject must plan to receive all 6 Radium Ra 223 dichloride injections and daily oral doses of Abiraterone plus Prednisone during the trial, per protocol.
8. Subject has a history of bone metastasis from prostate cancer as evidenced by imaging performed within 90 days of enrollment from one of the following:

   • Tc Bone Scan or

   • Sodium Fluoride PET/CT Scan

   *If a bone scan is used, solitary lesions which could be contributed to causes other than prostate cancer must be confirmed with a second modality (i.e.: plain films, CT Scan or MRI.
9. Subject has Castrate Resistant Prostate Cancer, defined as rising PSA with a testosterone level </= 50ng/dl (2.0 nM/L) while receiving androgen deprivation therapy (medical or surgical castration).

   * PSA progression will be defined as at least 2 rising PSA levels taken at least 7 days apart with the 2nd PSA being 2.0 ng/dl or greater.
10. Subject has the presence of bone pain requiring treatment with:

1) EBRT within the previous 12 weeks prior to enrollment, or 2) Analgesic medications (including but not limited to acetaminophen, NSAIDS, Cox-2 inhibitors, and narcotic Opioids).

11. Subject has an ECOG performance status of 0-2 at screening 12. Acceptable hematology and serum biochemistry screening values:

• White Blood Cell (WBC) >/= 3,000/mm3

* Absolute Neutrophil Count (ANC) >1500/mm3
* Platelet (PLT) count >100,000/mm3
* Hemoglobin (HGB) > 10.0 g/dL (100g/L; 6.2 mmol/L
* Creatinine <1.5 ULN
* Total bilirubin level <1.5 X ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 X ULN
* albumin >25 g/L
* Baseline electrolytes within normal limits ( Sodium, potassium, chloride, calcium, phosphate, magnesium, LDH, γGT, urea, total protein) 13. Normal Liver Function Tests (LFT) and normal Renal Function Tests (RFT) at screening visit. If the subject has LFT's or RFT's greater than 2.5 times the upper limit of normal (ULN), Medical Monitor review, in conjunction with the subject's PI, will be required.

  14. Subjects receiving Anti-Resorptive medications (such as Zolendronic Acid or denosumab) must be on a stable dose for at least 90 days prior to enrollment (Cycle 1/Week 1/ Day 1). Anti-resorptive medications may be added to the subject's regimen after the End of Treatment visit has been completed. Anti-resorptive medication withdrawal will be allowed per Investigator discretion due to adverse events attributable to that medication.

  15. Subjects of childbearing potential must agree to use adequate contraception beginning at the enrollment until at least 30 days after the last dose of the study drugs. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.

Exclusion Criteria:

Eligible subjects must not meet any of the exclusion criteria listed below:

1. Subject has known malignant pleural effusion, or known lung, liver or brain metastasis (lymph node only metastasis < 6 cm in short-axis diameter is allowed).
2. Subject has a history of visceral metastatic disease as assessed by abdominal/pelvic CT or chest x-ray within the previous 8 weeks.
3. Subject has received previous treatment with Abiraterone Acetate for longer than 90 days prior to enrollment, or any prior treatment with Radium Ra 223 dichloride.
4. Subject has a known medical contraindication to Prednisone, Abiraterone Acetate or Radium Ra 223 dichloride.
5. Subject is not willing to initiate a stable dose of daily Abiraterone Acetate plus Prednisone within 90 days of enrollment, or does not plan to initiate a stable daily dose of Abiraterone Acetate plus Prednisone within 30 days of the first Radium Ra 223 dichloride treatment.
6. Subject does not plan to receive all 6 infusions of Radium Ra 223 Dichloride and daily Abiraterone Acetate plus Prednisone during the trial, per protocol.
7. Subject has received previous strontium-89, samarium-153, rhenium-186, or rhenium-188 for the treatment of bone metastasis within 24 weeks prior to enrollment.
8. Subject has received denosumab or Zolendronic Acid for less than 90 days prior to enrollment, or if the subject plans to discontinue an anti-resorptive medication prior to the EOT visit.
9. Subject has received an investigational product or experimental therapy within 4 weeks of enrollment, or if initiation of either is planned prior to the EOT visit.
10. Subject has had treatment with cytotoxic chemotherapy within the previous 4 weeks, or planned prior to the End of Treatment visit, or failure to recover from adverse events due to cytotoxic chemotherapy administered more than 4 weeks prior to enrollment (persistent myelosuppression, GI toxicity, or severe fatigue (ongoing neuropathy is not exclusionary).
11. Subject has a history of any medical condition that may be compromised by an increase in blood pressure, or severe liver insufficiency (r Child-Pugh class B or C).
12. Subject has a history of a myocardial infarction or cardiac arrhythmia within 6 months prior to enrollment.
13. Subject has a history of previous radiotherapy >25% of bone marrow, including hemibody radiation.
14. Subject has a history of any other malignancy within the previous 5 years. A history of squamous or basal cell carcinoma or low-grade superficial bladder cancer that has been adequately treated at least 12 months prior to enrollment is not exclusionary.
15. Subject has undergone major surgery within 4 weeks prior to enrollment.
16. Subject has had a blood transfusion or erythropoietin stimulation agents within 4 weeks of enrollment.
17. Subject has known imminent or established spinal cord compression.
18. Subject has a serious concurrent medical condition or psychiatric illness.
19. Subject has a history of other serious illness of medical condition including, but not limited to any uncontrolled infection, congestive heart failure New York Heart Association (NYHA) class III or IV, Crohn's Disease or Ulcerative Colitis, uncontrolled hypertension or Bone Marrow Dysplasia at screening.
20. Subject has any condition that, in the opinion of the investigator, would impair the patient's ability to comply with study procedures.
21. Subject is not able to swallow the study treatment capsules.
22. Subject has unmanageable fecal incontinence.
23. Subject has a history of any size pelvic lymphadenopathy if it is thought to be a contributor to current hydronephrosis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Shore, MD, Principal Investigator — Carolina Research Professionals, LLC
Locations (5):
- United States (5):
  - Chesapeake urology Research Associates, Towson, Maryland
  - Urology Cancer Center and GU Research Network, Omaha, Nebraska
  - Associated Medical Professionals, Syracuse, New York
  - Oregon Urology Institute, Springfield, Oregon
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Radium 223 With Concomitant Abiraterone Acetate and Prednisone: Name of active ingredient Radium Ra 223 dichloride Dose 50 kBq/kg body weight Route of Administration Intravenous Duration of Treatment One injection every 4 weeks X 6 injections maximum.
  Name of active ingredient Abiraterone Acetate plus Prednisone Dose 1000 mg/day and 5 mg BID Route of Administration Oral Duration of Treatment 26 weeks minimum duration. There is no maximum duration.
Period: Overall Study
Arm/Group | Radium 223 With Concomitant Abiraterone Acetate and Prednisone
Started | 36
Completed | 31
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Radium 223 With Concomitant Abiraterone Acetate and Prednisone
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 75 [51 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic or Latino | 36
  Caucasian | 28
  African American | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Clinically Meaningful Improvement (Between Baseline and End of Treatment) in Quality-of-Life Determined by the Minimum Increase From Baseline in Scores as Per the QOL CMI Criteria
Description: Following Quality of Life questionnaires were given at each visit:
  FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the PCS (Range 1-156, higher scores better).
  The FACT-General (FACT-G) is a 28 item QOL measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), Emotional (0-24) Well-being, and Satisfaction with Treatment was not assessed for this study (The total range was between 1-108, higher scores better)
  FACT-TOI is derived from the sum of the Physical Well-Being, Functional Well-Being, and Prostate Cancer subscale scores; a sensitive measure of patient-reported health (Range 1-104, higher scores better)
  PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better).
Time Frame: Subjects were evaluated at the screening visit, monthly during the study, and 30 days after the last dose of Radium Ra 223 dichloride, which will be approximately 32 weeks after the screening visit of evaluable subjects.
Population: Improvement at the EOT visit was defined as increase from baseline of >= 10 points for FACT-P Total Scale. >9 points for FACT-G Total and FACT-TOI scales, and >=3 points for the remaining scales.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium 223 With Concomitant Abiraterone Acetate and Prednisone
Number analyzed (Participants) | 31
Participants
  FACT-P Total Scale | 20
  FACT-G Total Scale | 18
  Treatment Outcome Index (FACT-TOI) | 18
  Prostate Cancer Subscale (PCS) | 25
  Physical Well-being | 19
  Functional Well-being | 17
  Emotional Well-being | 18
  Social Well-being | 15

2. Secondary Outcome: Safety Data Was Analyzed and Summarized in Subjects Who Receive at Least One Infusion of Radium Ra 223 Dichloride. Number of Adverse Events Are Being Reported.
Description: All adverse events relevant to advanced mCRPC subjects as well as adverse events of interest for both Abiraterone Acetate plus Prednisone and Radium Ra 223 dichloride will be reported.
Time Frame: as for outcome 1
Measure: Number; unit: Adverse Events
Arm/Group | Radium 223 With Concomitant Abiraterone Acetate and Prednisone
Number analyzed (Participants) | 36
Adverse Events
  Overall Adverse Events | 186
  Grade I or II Adverse Events | 179
  Treatment Related Adverse Events | 70

3. Secondary Outcome: Alkaline Phosphatase (ALP) and Prostate Specific Antigen (PSA) Levels Before and After Treatment
Description: [Not specified]
Time Frame: Baseline and End of Treatment (EOT), approximately 32 weeks from Baseline
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Radium 223 With Concomitant Abiraterone Acetate and Prednisone
Number analyzed (Participants) | 31
ng/dL
  ALP (Baseline) | 261 (284)
  ALP (EOT) | 110 (187)
  PSA (Baseline) | 87 (233)
  PSA (EOT) | 137 (441)
Statistical Analysis 1: Comparison: Radium 223 With Concomitant Abiraterone Acetate and Prednisone; Test type: Other; p < .00001, t-test, 2 sided — Comparison of ALP levels before and after treatment
Statistical Analysis 2: Comparison: Radium 223 With Concomitant Abiraterone Acetate and Prednisone; Test type: Other; p = 0.4870, t-test, 2 sided — Comparison of PSA levels before and after treatment

4. Secondary Outcome: Radiologic Assessment Mean Number of Bone Lesions Before and After the Treatment
Description: [Not Specified]
Time Frame: Baseline and End of Treatment (EOT), approximately 32 weeks from Baseline
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Radium 223 With Concomitant Abiraterone Acetate and Prednisone
Number analyzed (Participants) | 31
Lesions
  Baseline | 11.6 (2.8)
  EOT | 5.6 (2.4)

5. Other Pre Specified Outcome: Bone Imaging Response (Number of Participants With Progression and Stable Disease)
Description: Bone imaging response was assessed at baseline and at EOT visit. Progression was defined as two or more additional lesions in comparison to the baseline.
Time Frame: Baseline and End of Treatment (EOT), approximately 32 weeks from Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Radium 223 With Concomitant Abiraterone Acetate and Prednisone
Number analyzed (Participants) | 31
Participants
  Stable Disease | 29
  Progression | 2

6. Primary Outcome: Number and Percentage of Participants With Clinically Meaningful Improvement (CMI) in Pain (Between Baseline and End of Treatment)
Description: Improvement in Bone Pain was assessed using the Bone Pain Inventory (BPI)
  1. Pain Severity: Pain severity is the composite of scores of worst pain, least pain, average pain, and pain now. CMI criteria: Decrease >30% at two consecutive visits in Pain Severity Score in 24 hours without an increase in analgesic use.
  2. Pain interference: Pain interference is the composite scores on general activity, mood, walking ability, normal work, relationships with others, sleep and enjoyment of life. CMI criteria: Decrease by 1.25 points or more compared with baseline at two consecutive visits.
  3. Transient Pain Flare: Based on the work of Atkinson et al, a transient pain flare was assessed by pain at its worst in 24 hours. CMI criteria: > 2 points on the BPI-SF Worst Pain scale and subsequent reduction after initiation of Ra-223 and during the first 3 cycles.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Radium 223 With Concomitant Abiraterone Acetate and Prednisone
Number analyzed (Participants) | 31
Participants
  Pain Severity | 18
  Pain Interference | 12
  Transient Pain Flare | 2

7. Other Pre Specified Outcome: Overall Response Rate
Description: Determination of measurable disease progression or response was based on modified RECIST criteria. Reported is the number of participants with either a partial or complete response, and who had radiological extraskeletal progression.
Time Frame: Baseline and End of Treatment (EOT), approximately 32 weeks from Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Radium 223 With Concomitant Abiraterone Acetate and Prednisone
Number analyzed (Participants) | 31
Participants
  Partial or complete response | 4
  Progression | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through 6 monthly cycles, and 30 days after the end of treatment, for a total of 7 months.
Arm/Group | Radium 223 With Concomitant Abiraterone Acetate and Prednisone
All-Cause Mortality (participants affected / at risk) | 1/36
Serious Adverse Events (participants affected / at risk) | 5/36
Other Adverse Events (participants affected / at risk) | 30/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium 223 With Concomitant Abiraterone Acetate and Prednisone (N=36)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Deemed treatment related.
Cardiopulmonary Arrest (Cardiac disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium 223 With Concomitant Abiraterone Acetate and Prednisone (N=36)
Anemia (Blood and lymphatic system disorders) | 5 (9)
Leukopenia (Blood and lymphatic system disorders) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 2 (4)
Pancytopenia (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 7 (14)
Nausea (Gastrointestinal disorders) | 7 (21)
Stomach Pain (Gastrointestinal disorders) | 2 (4)
Abdominal Pain (Gastrointestinal disorders) | 1 (2)
Decreased Appetitie (Gastrointestinal disorders) | 1 (3)
Dysguesia (Gastrointestinal disorders) | 1 (1)
Edema Limbs (Blood and lymphatic system disorders) | 3 (6)
Fatigue (Endocrine disorders) | 6 (14)
Increased Liver Function Tests (Hepatobiliary disorders) | 1 (3)
Decreased Red Blood Count (Blood and lymphatic system disorders) | 1 (3)
Increased ALT (Hepatobiliary disorders) | 2 (4)
Increased ALT (Hepatobiliary disorders) | 2 (5)
Increased ALP (Hepatobiliary disorders) | 1 (2)
Hypocalcemia (Investigations) | 2 (3)
Hyponatremia (Investigations) | 2 (4)
Hyponatremia (Investigations) | 1 (2)
Hypochloremia (Investigations) | 1 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3)
Dizziness (Ear and labyrinth disorders) | 2 (5)
Headaches (Ear and labyrinth disorders) | 1 (3)
Paresthesia (Ear and labyrinth disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No